CLINICAL TRIAL: NCT00550329
Title: An Open-Label, Randomized, Single-Dose, Two-Way Crossover Bioequivalence Study Of Glucotrol XL 2.5 Mg Tablets Manufactured At Brooklyn, New York Versus At Barceloneta, Puerto Rico In Healthy Subjects
Brief Title: Bioequivalence Study Of Glucotrol XL 2.5 Mg Tablets
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Other Study IDs: A1251009
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Glipizide GITS

SUMMARY:
The objective of this study is to determine the bioequivalence of Glipizide GITS (Glucotrol XL) 2.5 mg tablets manufactured at the Brooklyn, New York facility versus tablets manufactured at the facility in Barceloneta, Puerto Rico.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests). Subjects below the age of 21 years must have consent from either a parent or guardian in countries having this requirement.
2. Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >45 kg (99 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
4. Subjects who are willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Any condition possibly affecting drug absorption (e.g., gastrectomy).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
5. History or evidence of habitual tobacco- or nicotine-containing products within 3 months of screening or a positive urine or serum cotinine test.
6. Treatment with an investigational drug within 30 days preceding the first dose of study medication.
7. 12-lead ECG demonstrating QTc >450 msec at Screening.
8. Sitting blood pressure ?140 mm Hg systolic or ?90 mm Hg diastolic on a single measurement [confirmed by a single repeat, if necessary] following at least 5 minutes of rest at Screening.
9. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication until completion of follow-up procedures.
10. Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. Depo-Provera� must be discontinued at least 6 months prior to the first dose of study medication. As an exception, acetaminophen may be used at doses of ?1g/day. Other exceptions may be granted by a qualified member of Pfizer study management.
11. Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
12. Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2007-10; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1251009&StudyName=Bioequivalence%20Study%20Of%20Glucotrol%20XL%202.5%20Mg%20Tablets